CLINICAL TRIAL: NCT05301127
Title: Combination of Spinal-Epidural With General Anesthesia in Patients Undergoing Mega-Liposuction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-54-2021
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Combination of General Anesthesia to Spinal and Epidural Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSEGA group (Active Comparator): Will be received combined spinal-epidural-general anesthesia.
  Interventions: Device: spinal-epidural device
- GA group (No Intervention): will be received general anesthesia only.

INTERVENTIONS:
Device: spinal-epidural device — received combined spinal-epidural-general anesthesia.
  Arms: CSEGA group

SUMMARY:
The combination of general anesthesia to spinal and epidural techniques (CSEGA) proved to have a synergistic effect, thus, the use of sub-anesthetic doses can provide satisfactory anesthetic and analgesic results. CSEGA has several known advantages including appropriate postoperative analgesia, shows some benefit in the intraoperative blood loss control causing a decreased need for blood transfusion, rapid regain of the gastrointestinal actions and decreases the incidence of postoperative respiratory complications. Unfortunately, the drawbacks of using neuro-axial anesthesia in combination to general anesthesia will be not thoroughly introduced in many researches, thus, remain unclear.

ELIGIBILITY:
1. Inclusion criteria:

   * Patients aged from 18 to50 years.
   * ASA I-II.
   * undergoing elective liposuction surgery
   * BMI from 25 to 40 kg/m2
2. Exclusion criteria:

   * Patient refusal
   * ASA III-IV.
   * Patients aged less than 18 or more than 50.
   * Body mass index >40.
   * Any contraindications to neuro-axial block such as coagulopathy or spine deformity
   * Chronic opioid consumption,
   * History of parenteral or oral analgesic intake within the last 48hours.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  postoperative morphine consumption

SECONDARY OUTCOMES:
Postoperative patient satisfaction | 24 hours
  1 = very unsatisfactory; 2 = unsatisfactory; 3 = indifferent; 4 = satisfactory; and 5 = very satisfactory.
Intraoperative surgeon satisfaction. | 6 hours
  using 1-4 scales (1, bad; 2, moderate; 3, good; 4, excellent;
Incidence of complications | 24 hours
  such as hypotension, bradycardia, nausea and vomiting, postoperative shivering,
Blood loss | 6 hours
  intraoperative Blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working